CLINICAL TRIAL: NCT00369460
Title: Pilot Study of Changes in Fat-Free Mass in Pancreatic Carcinoma Patients
Brief Title: Changes in Muscle Tissue in Patients With Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE8205; P30CA043703 (NIH); CASE8205 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: physiologic testing — Weight, body mass index, age, ECOG performance status, gait speed, concomitant medications, CA19-9, and total lymphocyte count measured before start of cancer treatment of the patient's choosing. Patients will be re-assessed at approximately 2 months, 4 months, 6 months, and with any change in tumor burden.

SUMMARY:
RATIONALE: Measuring changes in muscle tissue in patients with cancer may help doctors predict how well patients will respond to treatment, and may help the study of cancer in the future.

PURPOSE: This pilot study is evaluating changes in muscle tissue in patients with pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Demonstrate a decrease/increase of fat-free mass (FFM) by 10% from baseline, based on tumor progression/regression, within each patient with inoperable locally advanced or metastatic pancreatic carcinoma.
* Determine the correlation between changes in FFM and 6-month survival.
* Confirm the frequency of lymphocytopenia in patients with inoperable locally advanced or metastatic pancreatic carcinoma.
* Demonstrate an interaction between pretreatment total lymphocyte count, treatment response, and 6-month survival in patients with inoperable locally advanced or metastatic pancreatic carcinoma.
* Collect adjuvant information, such as weight, body mass index, age, ECOG performance status, gait speed, concomitant medications, CA19-9, and total lymphocyte count, in these patients.

OUTLINE: This is a pilot study.

Patients will have weight, body mass index, age, ECOG performance status, gait speed, concomitant medications, CA19-9, and total lymphocyte count measured before start of cancer treatment of the patient's choosing.

Patients will be re-assessed at approximately 2 months, 4 months, 6 months, and with any change in tumor burden.

PROJECTED ACCRUAL: A total of 17 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven inoperable locally advanced or metastatic pancreatic adenocarcinoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Must be able to stand unassisted on a scale
* Must not have pacemaker or implanted defibrillator

PRIOR CONCURRENT THERAPY:

* Prior chemotherapy or radiotherapy allowed
* No concurrent use of any of the following:

  * Corticosteroids

    * Steroids as anti-emetics associated with chemotherapy allowed
  * Anabolic steroids
  * Thalidomide
  * Megesterol
  * Eicosapentaenoic acid (EPA)

    * Nutritional supplements without EPA allowed
  * Juven
* Concurrent enrollment in other clinical trials allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Fat-free mass (FFM) | Patients will have body mass index measured before start of cancer treatment of the patient's choosing. Patients will be re-assessed at approximately 2 months, 4 months, 6 months, and with any change in tumor burden.
Correlation of changes in FFM with survival at 6 months | at 6 months
Incidence of lymphocytopenia | Total lymphocyte count measured before start of cancer treatment and at approximately 2 months, 4 months, 6 months, and with any change in tumor burden.
Correlation of pretreatment total lymphocyte count, treatment response, and survival at 6 months | at 6 months
Collection of information on weight, body mass index, age, ECOG performance status, gait speed, concomitant medications, CA19-9, and total lymphocyte count | At start of cancer treatment and re-assessed at approximately 2 months, 4 months, 6 months, and with any change in tumor burden.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M. Brell, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States